CLINICAL TRIAL: NCT02252224
Title: Post-Marketing Surveillance to Evaluate the Safety and Efficacy of Forxiga in Patients With Type 2 Diabetes in Korea
Brief Title: Forxiga (Dapagliflozin) Regulatory Postmarketing Surveillance
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690L00018
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- T2DM patients treated with Forxiga: Korean patients who are at least 18 years old, diagnosed with type2 diabetes and treated with Forxiga according to the approved lable

SUMMARY:
This surveillance is a postmarketing commitment following the marketing authorization for Forxiga(dapagliflozin) in accordance with Standards on Re-examination of New Drugs, notified by the MFDS under Article 32, Paragraph 1 and Article 37, Paragraph 3 of Pharmaceutical Affairs Law. MFDS requires that at least 3,000 patients who can be evaluated for safety assessment should be collected within 6 years from 26 Nov 2013 to 25 Nov 2019.

DETAILED DESCRIPTION:
Protocol Title: Forxiga (dapagliflozin) Regulatory Postmarketing Surveillance

Department: Korea Medical

Objective(s): The primary objective of this study is to examine the safety profiles of Forxiga in Korean patients with T2DM.

The secondary objective of this study is to examine the effectiveness profiles of Forxiga in Korean patient with T2DM.

The exploratory objective of this study is to identify factors that might be associated with the safety and effectiveness profiles of Forxiga in Korean patient with T2DM.

Study Design: This is a local, prospective, noninterventional, regulatory postmarketing surveillance study. Adult patients with type 2 diabetes mellitus who are initiating Forxiga as indicated by the Ministry of Food and Drug Safety (MFDS) will be included. Patients will be followed for a minimum of 12 weeks or a minimum 24 weeks. Patients will be treated as part of routine practice at Korean healthcare centers by accredited physicians. In this study, patients will receive 10 mg or 5 mg of Forxiga in conjunction with diet and exercise modifications for the treatment of T2DM.

Study Population: Physicians should enroll adult patients who are diagnosed with T2DM and who initiate treatment with 10 mg of Forxiga, or 5 mg of Forxiga in patients with severe hepatic impairment as a starting dose, for the first time.

Data Collection Methods: and Astra-Zeneca will select medical institutions including relevant departments, such as internal medicine and family medicine, of university hospitals, general hospitals and clinics where the surveillance drug is mainly prescribed and where staff can sufficiently fulfill the objectives of the surveillance and request for surveillance after signing a written contract. Patients' medical records will be data sources in this study. Only if the laboratory test is done as part of standard of care practice and the data are available will the data be collected for this study.

Data Analyses: Statistical analyses will be of explorative and descriptive nature. All analyses will be performed for the total study population who will consist of all patients taking at least one dose of Forxiga. For the safety assessment, occurrences of adverse events (AEs), serious adverse events, adverse drug reactions (ADR), and unexpected adverse drug reactions will be calculated. Severity, actions taken to the surveillance drug, outcome, and causal relationship of AE to the study drug will be analyzed. At the time of the regular reporting and the final reporting, the event count, incidence proportion (that is, the number of patients with any events divided by the number of patients) and incidence rate (number of patients with any events divided by the duration of time patients are followed up in the study) of all the adverse events surveyed during the re-examination period will be summarized, and 95% confidence interval will be presented. Changes in Hemoglobin A1c(HbA1c), Fasting plasma glucose(FPG), and Post-prandial glucose-2 hour(2-hr PPG) before and after administration of Forxiga will be analyzed. At the time of the regular reporting and the final reporting, the event count and effectiveness rate of improvement of lab result (HbA1c, FPG, and PPG), surveyed during the re-examination period will be summarized, and 95% confidence interval will be presented. In order to explore the factors that might influence safety and effectiveness profiles, the cumulative incidence proportion of adverse events and effectiveness rate will be analyzed by patients' background characteristics Sample Size/Power: In accordance with the guidelines provided by the MFDS, at least 3,000 patients will be enrolled. For the overall study population of approximately 3000 patients, the incidence proportion of infrequent adverse events(for example, an incidence proportion of 0.1%) can be estimated with a 95% CI of (0.02, 0.29) (n=3 patients with events).

Limitations/Strengths: The surveillance, with characteristics of a noninterventional, observation study, has no control group and will follow patients in usual clinical practice. Given these conditions, the types of safety and effectiveness data available for collection may be limited compared with other noninterventional clinical trials. This surveillance study will generate results from a wider range of data than those previously derived from the more limited clinical trial setting and will allow for longer follow up among a more varied patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients with T2DM eligible for treatment with Forxiga as indicated in the locally approved prescribing information
* Patients with evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients treated with Forxiga outside of the locally approved label in Korea
* Patients with contraindications for the use of Forxiga (as described in the Korean product label)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with type 2 diabetes mellitus who are initiating Forxiga
Sampling Method: Non-Probability Sample
Enrollment: 3123 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
The number and incidence rate of adverse events and serious adverse event including unexpected adverse drug reactions | Adverse event will be collected from baseline(Day1) to 3 days after 12 weeks (maximum 16 weeks) or 24 weeks (maximum 30 weeks))
  All patients should be evaluated if they received at least one dose of the study medication. Safety will be evaluated through: • Incidence of serious adverse events • Incidence of unexpected adverse drug reactions • Identification of AE profile in usual practice • Report of AE in routine office visit or through phone or e-mail follow up • Incidence of nonserious adverse events All AEs that occurred on the surveillance drug treatment or within 3 days after the end of the treatment, whether or not related to the drug, will be recorded. The safety assessment should include all undesirable changes of medical findings (including a clinical test finding) noted during medical visits as needed according to local practice guidelines and all AEs associated with surveillance drug administration.

SECONDARY OUTCOMES:
Changes in HbA1c before and after administration of Forxiga | Baseline, 12 weeks (maximum 16 weeks), 24 weeks (maximum 30 weeks) in case of long-term surveillance
  Medical records and laboratory test results will be used to determine effectiveness as judged by the investigator. Changes from baseline to at least 12 weeks (maximum 16 weeks) or 24 weeks (maximum 30 weeks) in case of long-term surveillance will be assessed for the following outcome measure (if assessed during routine clinical practice): HbA1c (Hemoglobin A1c)
Changes in FPG before and after administration of Forxiga | Baseline, 12 weeks (maximum 16 weeks), 24 weeks (maximum 30 weeks) in case of long-term surveillance
  Medical records and laboratory test results will be used to determine effectiveness as judged by the investigator. Changes from baseline to at least 12 weeks (maximum 16 weeks) or 24 weeks (maximum 30 weeks) in case of long-term surveillance will be assessed for the following outcome measure (if assessed during routine clinical practice): FPG (fasting plasma glucose)
Changes in 2-hr PPG before and after administration of Forxiga | Baseline, 12 weeks (maximum 16 weeks), 24 weeks (maximum 30 weeks) in case of long-term surveillance
  Medical records and laboratory test results will be used to determine effectiveness as judged by the investigator. Changes from baseline to at least 12 weeks (maximum 16 weeks) or 24 weeks (maximum 30 weeks) in case of long-term surveillance will be assessed for the following outcome measure (if assessed during routine clinical practice): 2-hr PPG (2-hr post-prandial glucose)

CONTACTS AND LOCATIONS:
Overall Officials: A Ri Kim, Study Director — AstraZeneca Korea - Medical Affairs
Locations (6):
- South Korea (6):
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Daejeon
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Wŏnju

REFERENCES:
- [Derived] Han E, Kim A, Lee SJ, Kim JY, Kim JH, Lee WJ, Lee BW. Characteristics of Dapagliflozin Responders: A Longitudinal, Prospective, Nationwide Dapagliflozin Surveillance Study in Korea. Diabetes Ther. 2018 Aug;9(4):1689-1701. doi: 10.1007/s13300-018-0470-9. Epub 2018 Jul 11. PMID 29998370